CLINICAL TRIAL: NCT07070856
Title: Efficacy and Safety of Therapeutic Rice Based F75 In Severely Acute Malnourished Children With Persistent Diarrhea.;A Randomized Control Trial.
Brief Title: Trial of Rice-Based F-75 in Severe Malnutrition & Persistent Diarrhea in Children (SAM-RICE Study)
Acronym: SAM-RICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital and Institute of Child Health, Multan (Other Government)
Responsible Party: Principal Investigator, Dr. Saadia Khan, Pricipal Investigator, Children's Hospital and Institute of Child Health, Multan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1324-6540
Record Dates: First submitted 2025-06-28; First posted 2025-07-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Severe Acute Malnutrition; Persistent Diarrhea; Children
Keywords: Severe Acute Malnutrition; Persistent Diarrhea; F-75 Formula; Rice-Based Diet; Nutritional Rehabilitation; Protein-Energy Malnutrition; Lactose intolerance
MeSH Terms: conditions — Severe Acute Malnutrition; Protein-Energy Malnutrition; Lactose Intolerance | interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHO standard f75 (Active Comparator): standard ,prepared.powdered F75 by WHO
  Interventions: Dietary Supplement: WHO-recommended standard therapeutic milk used for stabilization phase in SAM)
- Rice Based F75 (Experimental): Rice based F75 BY WHO recipe for PERSISTENT Diarhea
  Interventions: Dietary Supplement: HO-recommended Rice based therapeutic milk used for stabilization phase in SAM)

INTERVENTIONS:
Dietary Supplement: WHO-recommended standard therapeutic milk used for stabilization phase in SAM) — F75 GIVEN INITIALLY 2HOURLY,130 ml per kg than 3 and 4hourly maximum takes 5 to 7 days.
  Other Names: Stabalization phase feed
  Arms: WHO standard f75
Dietary Supplement: HO-recommended Rice based therapeutic milk used for stabilization phase in SAM) — Rice based F75 GIVEN INITIALLY 2HOURLY,130 ml per kg than 3 and 4hourly maximum takes 5 to 7 days.
  Arms: Rice Based F75

SUMMARY:
The goal of this study is to find out if a rice-based version of the F-75 therapeutic food helps children with severe acute malnutrition (SAM) and persistent diarrhea recover better than the standard commercial F-75.

The main questions it aims to answer are:

1. Does rice-based F-75 reduce the duration of diarrhea and improve nutritional recovery in children with SAM?
2. Is rice-based F-75 as safe and well-tolerated as the standard WHO F-75?

Researchers will compare two groups:

One group will receive the new rice-based F-75. The other group will receive the standard F-75.

Participants will:

1. Be children aged 6 to 59 months admitted with SAM and persistent diarrhea
2. Be randomly assigned to one of the two feeding groups
3. Stay in a hospital ward for monitoring during the stabilization phase

Be assessed daily for:

Stool frequency Weight changes Appetite Medical problems or side effects

This study will help determine whether the rice-based F-75 is a better option for malnourished children with diarrhea.

DETAILED DESCRIPTION:
Persistent diarrhea in children with severe acute malnutrition (SAM) poses a significant clinical challenge, particularly during the stabilization phase. Standard therapeutic protocols include the use of F-75-a milk-based formula designed to meet the reduced metabolic demands of severely malnourished children. However, lactose content in milk-based F-75 may exacerbate intestinal symptoms in children with secondary lactase deficiency, commonly observed in cases of persistent diarrhea.

Rice-based therapeutic formulations have emerged as promising alternatives, potentially offering superior gastrointestinal tolerance, improved nutrient absorption, and reduced osmolarity compared to conventional milk-based F-75. Rice is hypoallergenic, low in anti-nutritional factors, and contains resistant starches that may support gut integrity and microbial balance during intestinal recovery.

Introducing rice-based F-75 may address dietary intolerance in children with diarrhea-induced lactase deficiency, particularly in low-resource settings where commercial lactose-free preparations are unavailable or unaffordable. This trial seeks to assess whether therapeutic feeding with rice-based F-75 leads to faster stabilization without compromising metabolic safety or nutritional adequacy.Participants are randomized into intervention and control arms during hospitalization, receiving either rice-based or conventional F-75 during the stabilization phase. Transition to F-100 occurs per clinical criteria once acute symptoms resolve.

Clinical monitoring includes:

* Gastrointestinal Tolerance: Stool frequency, consistency, abdominal distension, emesis, and need for additional rehydration.
* Metabolic Safety: Serum sodium, potassium, bicarbonate, and creatinine levels evaluated at baseline and mid-stabilization.
* Nutritional Stabilization: Daily weight, mid-upper arm circumference (MUAC), and feeding tolerance.
* Adverse Events Surveillance: Identification of allergic responses, metabolic complications, or mortality.

ELIGIBILITY:
Inclusion Criteria:

* All the children admitted to the hospital with complaints of persistent diarrhea
* secondary lactose

Exclusion Criteria:

* All the children with primary lactose intolerance
* Those parents /guardians refused permission to participate in the study.
* Critically ill child admitted to ICUs and emergency department.
* Patients started therapeutic feeding prior to recruitment in study .

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
stool frequency | day 1 to day 7 of starting therapeutic feed
  episodes of loose stools per day

OTHER OUTCOMES:
hydration status | day 1 to day 7 of treatment
  IMNCI Protocol
Re feeding syndrome | Day 1 to day 7 of treatment with therapeutic feed
  monitoring of vitals,edema,heart failure,electrolytes imbalance,convulsions
Electrolytes monitoring | Time Frame: Baseline and Day 4
  - Serum Sodium and potassium Unit of Measure: mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad T Sultan, PhD, Study Chair — Bahauddin zakariya University,Multan
Locations (2):
- Pakistan (2):
  - Tehsil Head Quater Sujah Abad, Multan Khurd, Punjab Province
  - The Childrens Hospital and Instotute of Child Health Multan, Multan Khurd, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Facioni MS, Raspini B, Pivari F, Dogliotti E, Cena H. Nutritional management of lactose intolerance: the importance of diet and food labelling. J Transl Med. 2020 Jun 26;18(1):260. doi: 10.1186/s12967-020-02429-2. PMID 32590986